CLINICAL TRIAL: NCT04145284
Title: Performance and Feasibility of Quantitative MRI Metrics in Routine Radiology Practice: A Sub-Study of MS PATHS
Brief Title: Quantitative Magnetic Resonance Imaging (MRI) Sub-Study of MS PATHS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 888MS007
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to assess the performance of a new magnetic resonance imaging (MRI) metrics software prototype when used in radiological practice in multiple sclerosis (MS).

ELIGIBILITY:
Key Inclusion Criteria:

* Board-certified neuroradiologists or experienced neuroradiology fellows.
* Employed at a participating MS PATHS institution.
* At least 3 years of experience in interpreting brain MRI scans of MS participants.

Key Exclusion Criteria:

* Inability to comply with sub-study procedures.
* Other unspecified reasons that, in the opinion of Biogen or the MS PATHS Radiology Lead at the institution, make the radiologist unsuitable for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the cohort of radiologists.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Radiologist Assessment of the Performance of the MS MRI Metrics Software Prototype by the Number of Approve or Reject Decision | Baseline up to 6 weeks
  MRIs from participants will be analyzed by the prototype. The radiologist will view the brain segmentation results and the new or enlarging T2 lesion detection results. The radiologist will either "Approve" or "Reject" the results.
Radiologist Assessment of the Performance of the MS MRI Metrics Software Prototype by the Number of False-Positive and False-Negative Lesions | Baseline up to 6 weeks
  MRIs from participants will be analyzed by the prototype. The radiologist will view the new or enlarging T2 lesions to determine false-positive or false-negative results.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- Research Site, Cleveland, Ohio, United States
- Research Site, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/